CLINICAL TRIAL: NCT03981133
Title: The Missing Answer: When is it Safe to Introduce the Pacifier to the Breastfed Baby? A Multicenter, Randomized, Control Trial
Brief Title: Influence of Unrestricted Introduction of Pacifiers on Breastfeeding Duration
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fundación para el Estudio y Prevención de la Muerte Infantil y Perinatal (Other)
Collaborators: Hospital Italiano de Buenos Aires (Other); Fundacion para la Salud Materno Infantil (Other)
Responsible Party: Principal Investigator, Alejandro Jenik, Professor consultant pediatrics, Fundación para el Estudio y Prevención de la Muerte Infantil y Perinatal
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: marita909
Record Dates: First submitted 2019-06-06; First posted 2019-06-10 (Actual); Last update posted 2019-06-10 (Actual); Status verified 2019-06

CONDITIONS: Lactation
Keywords: pacifier; breastfeeding; sudden unexpected infant death
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A: unrestricted pacifier (Experimental): recommendation to offer a pacifier at the facility providing maternity and newborn services the first days of life
  Interventions: Behavioral: offer a pacifier
- restricted pacifierr (Active Comparator): recommendation not to offer a pacifier to normal new born infant at the maternity thre first days of live
  Interventions: Behavioral: no pacifier

INTERVENTIONS:
Behavioral: offer a pacifier — offer a pacifier to normal newborn infants the first days of life
  Arms: A: unrestricted pacifier
Behavioral: no pacifier — not to offer a pacifier at 15 days of life
  Arms: restricted pacifierr

SUMMARY:
We will enroll 1010 mother-infant dyads in a randomized trial exploring the effect of distribution of the pacifier during the first days of life on breastfeeding prevalence and duration. .

DETAILED DESCRIPTION:
Given the scarcity of scientifically rigorous studies that address the impact of unrestricted pacifier exposure on breastfeeding we plan to conduct a multicenter, randomized, single blind, active control, parallel assignment, efficacy study to assess the impact of offering a pacifier on breastfeeding during the first days of life our hypothesis is that the introduction of a pacifier during the first days of life does not interfere with lactation

A research assistant will approach all eligible mothers during the first 6 hours after birth and will invite them to be randomized to one of the two groups:

Unrestricted pacifier ( the pacifiers can be offered liberally to infants to suck on during their stay at the facility providing maternity and newborn services) and Restricted pacifier group: ( avoid pacifier use until breastfeeding is well established) Women will be followed up at 1, 3, 4, ,6, 8, and 12 months after birth or until breastfeeding ended by a research assistant blinded to the group assignment. Interviews will be conducted by telephone using structured questionnaires designed to assess breastfeeding (exclusive or partial) prevalence and duration, and whether or not the baby had rejected a pacifier the night before the telephone interview. Rates of exclusive, partial, and any other occasional random breastfeeding will be tracked at all these time points.

ELIGIBILITY:
Inclusion Criteria

* Understands the benefits and risk for offer liberally the pacifier during their stay at the maternity.
* Expressed an intention to breast feed exclusively their infant for at least 3 -months
* Possibility of contact by telephone
* Has the decision to offer a pacifier to the newborn infant , but not definite opinion about when are going to offer a pacifier
* Primiparous single birth
* Mother´s age 18 years or more

Exclusion Criteria:

* Maternal risk factors for lactation

  * Lack of noticeable breast enlargement during pregnancy
  * Flat or inverted nipples
  * Variation in breast appearance (marked asymmetry, hypoplastic, tubular)
  * Any previous breast surgery, including plastics procedure
* Psychosocial problems (eg, depression, poor or negative support of breastfeeding
* Mother with a chronic condition that could influence development , including feeding ability
* Mother with eating or mental disorder.
* Mothers who smoke during pregnancy

Ages: 6 Hours to 3 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1010 (Estimated)
Dates: Start 2020-01 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Prevalence of exclusive breastfeeding | up to 24 weeks
  To compare the prevalence of exclusive breastfeeding at three, four and six months in infants between groups randomized to unrestricted pacifier group and restricted pacifier group

SECONDARY OUTCOMES:
infant feeding - breastfeeding duration | up to 24 weeks
  to evaluate the duration of exclusive and any breastfeeding duration in months between the two groups

CONTACTS AND LOCATIONS:
Overall Officials: alejandro G Jenik, MD, Principal Investigator — Fundacion para el Estudio y la Prevencion de la Muerte Infantil y Perinatal; Aleajndro G Jenik, MD, Principal Investigator — Fundacion para erl Estudio y Prevencionde la Muerte Subita y Perinatal
Locations (6):
- Argentina (6):
  - Hospital Privado de del Sur, Bahía Blanca, Buenos Aires
  - Hospital Italiano de buenos Aires, CABA, Buenos Aires
  - Sanatorio de la Trinidad, CABA, Buenos Aires
  - Alejandro Jenik, Olivos, Buenos Aires
  - Hospital Municipal Materno Infantil de San Isidro "Dr. Carlos Gianantonio"t, San Isidro, Buenos Aires
  - Centro Agustin Rocca HIBA, San Justo, Buenos Aires

IPD SHARING:
Plan to Share IPD: Yes
weight,gestational age,mother age, vaginal, cesarean,bedsharing, contact skin to skin
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: data will be available within 6 months of study
Access Criteria: data access requests will be reviewed by an external independent review panel. Requestors will be required to sifn a Data Access Agreement
URL: http://sids.org.ar